CLINICAL TRIAL: NCT01424137
Title: Inspiratory Flow Parameters With Placebo Dry Powder Inhalers, Easyhaler and Diskus; an Open, Randomised, Multicentre Study in Patients With Asthma or COPD
Brief Title: Inspiratory Flow Parameters of Easyhaler and Diskus Inhalers (SALIF)
Acronym: SALIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3106002
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Easyhaler type A (Other)
  Interventions: Device: Easyhaler type A
- Easyhaler type B (Other)
  Interventions: Device: Easyhaler type B
- Diskus inhaler (Other)
  Interventions: Device: Diskus inhaler

INTERVENTIONS:
Device: Easyhaler type A — Easyhaler type A inhaler, 3 consecutive inhalations
  Other Names: SF EH (D94-2SF)
  Arms: Easyhaler type A
Device: Easyhaler type B — Easyhaler type B inhaler, 3 consecutive inhalations
  Other Names: SF EH (D94-2SF-B)
  Arms: Easyhaler type B
Device: Diskus inhaler — Diskus inhaler, 3 consecutive inhalations
  Other Names: Inhaler for Seretide Diskus
  Arms: Diskus inhaler

SUMMARY:
The purpose of this study is to characterise inspiratory flow parameters across 2 Easyhaler® (EH) inhaler versions and Diskus® inhaler in patients with asthma (including children, adults, and the elderly) and in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained
* Documented diagnosis of asthma and/or COPD
* Age: 4 years and above

Exclusion Criteria:

* Any severe chronic respiratory disease other than asthma or COPD
* Acute respiratory infection
* Any medical condition that in the opinion of the investigator would endanger the subject if he/she participates in the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Peak inspiratory flow rate through the placebo Easyhaler and Diskus inhalers | 1 day

SECONDARY OUTCOMES:
The inspiratory volume through the placebo Easyhaler and Diskus inhalers will be measured at the same time with the peak inspiratory flow rate | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kati Kaijasilta, Study Director — Orion Corporation, Orion Pharma
Locations (5):
- Estonia (3):
  - Lasnamäe Medicum, Tallinn
  - Children's Clinic of Tartu, Allergy Centre, Tartu
  - Tartu University Hospital, Lung Clinic, Tartu
- Finland (2):
  - Jorvi Hospital HUS, Espoo
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Kainu A, Vartiainen VA, Mazur W, Hisinger-Molkanen H, Lavorini F, Janson C, Andersson M. Successful Use of Easyhaler(R) Dry Powder Inhaler in Patients with Chronic Obstructive Pulmonary Disease; Analysis of Peak Inspiratory Flow from Three Clinical Trials. Pulm Ther. 2024 Mar;10(1):133-142. doi: 10.1007/s41030-023-00246-8. Epub 2024 Jan 3. PMID 38170393